CLINICAL TRIAL: NCT04318002
Title: A Phase Ib Clinical Trial to Assess the Safety and Immunogenicity of the Blood-stage Plasmodium Falciparum Malaria Vaccine Candidate RH5.1/Matrix-M in Healthy Adults and Infants in Tanzania
Brief Title: Safety and Immunogenicity of RH5.1/Matrix-M in Adults and Infants Living in Tanzania
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Ifakara Health Institute (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: VAC080
Record Dates: First submitted 2020-02-13; First posted 2020-03-23 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2023-09

CONDITIONS: Malaria,Falciparum
Keywords: Vaccine
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1A (Experimental): Volunteers (aged 18-45 years) of low malaria exposure status will receive 3 doses of 10µg RH5.1 /50µg Matrix-M intramuscularly at months 0, 1 and 2
  Interventions: Biological: RH5.1/Matrix-M
- Group 1B (Experimental): Volunteers (aged 18-45 years) of low malaria exposure status will receive 2 doses of 50µg RH5.1 /50µg Matrix-M intramuscularly at months 0, 1 and 1 dose of 10µg RH5.1 /50µg Matrix-M at month 6.
  Interventions: Biological: RH5.1/Matrix-M
- Group 2A (Experimental): Volunteers (aged 5-17 months) of low malaria exposure status will receive 3 doses of 10µg RH5.1 /50µg Matrix-M intramuscularly at months 0, 1 and 2.
  Interventions: Biological: RH5.1/Matrix-M
- Group 2B (Experimental): Volunteers (aged 5-17 months) of low malaria exposure status will receive 3 doses of 10µg RH5.1 /50µg Matrix-M intramuscularly at months 0, 1 and 6.
  Interventions: Biological: RH5.1/Matrix-M
- Group 2C (Experimental): Volunteers (aged 5-17 months) of low malaria exposure status will receive 2 doses of 50µg RH5.1 /50µg Matrix-M intramuscularly at months 0, 1 and 1 dose of 10µg RH5.1 /50µg Matrix-M at month 6.
  Interventions: Biological: RH5.1/Matrix-M
- Group 2D (Experimental): Volunteers (aged 5-17 months) of high malaria exposure status will receive 2 doses of 50µg RH5.1 /50µg Matrix-M intramuscularly at months 0, 1 and 1 dose of 10µg RH5.1 /50µg Matrix-M at month 6.
  Interventions: Biological: RH5.1/Matrix-M

INTERVENTIONS:
Biological: RH5.1/Matrix-M — 3 doses of RH5.1/Matrix-M at different concentrations: RH5.1(10µg)/Matrix-M (50µg), RH5.1(50µg)/ Matrix-M (50µg), RH5.1(10µg)/ Matrix-M (25µg), RH5.1(50µg)/ Matrix-M (25µg)

SUMMARY:
This is an age de-escalation, dose-escalation open label randomised trial studying the safety and immunogenicity of RH5.1/Matrix-M, administered intramuscularly in healthy adults, young children and infants in Tanzania

DETAILED DESCRIPTION:
A total of 60 participants will be enrolled consisting of healthy adults (18-45 years) and infants (5-17 months) residing in Bagamoyo district, Tanzania. Participants will be recruited from areas of low malaria transmission in Bagamoyo town and areas of high malaria transmission within Bagamoyo district. All participants will be followed for 2-2.5years after the first vaccination with RH5.1/Matrix-M vaccination. The duration of the entire study will be 2-2.5years per participant from the time of first vaccination.

The trial is funded by EDCTP (reference: RIA2016V-1649 MMVC).

The paper containing this trial's results is available at: https://www.thelancet.com/journals/laninf/article/PIIS1473-3099(24)00312-8/fulltext

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Healthy male or female adults aged 18-45 years at the time of enrolment with signed consent.
* Group 1 (Female only participants): Must be non-pregnant (as demonstrated by a negative urine pregnancy test), and practice continuous effective contraception* for the duration of the study. (Female volunteers are required to use an effective form of contraception during the course of the study as this is a Phase I, study and there is currently no information about the effect of this vaccine on a foetus. Acceptable forms of contraception for female volunteers include:
* Established use of oral, injected or implanted hormonal methods of contraception.
* Placement of an intrauterine device (IUD) or intrauterine system (IUS).
* Total abdominal hysterectomy.
* Groups 2a, 2b, 2c & 2d: Healthy male or female infants aged 5-17 months at the time of enrolment with signed consent obtained from parents or guardians.
* Planned long-term (at least 24 months from the date of recruitment) or permanent residence in the study area.
* Adults with a Body Mass Index (BMI) 18 to 30 Kg/m2; or infants with Z-score of weight- for-age within ±2SD.

Exclusion Criteria:

* Clinically significant congenital abnormalities as judged by the PI or other delegated individual.
* Clinically significant history of skin disorder (psoriasis, contact dermatitis etc.), allergy, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease and neurological illness as judged by the PI or other delegated individual.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* Weight for age z-scores below 2 standard deviations of normal for age.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, e.g. egg products, Kathon, neomycin, betapropiolactone.
* Any history of anaphylaxis in relation to vaccination.
* Clinically significant laboratory abnormality as judged by the PI or other delegated individual.
* Blood transfusion within one month of enrolment.
* History of vaccination with previous experimental malaria vaccines.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period.
* Seropositive for hepatitis B surface antigen (HBsAg) or hepatitis C (HCV IgG).
* Any other finding which in the opinion of the PI or other delegated individual would increase the risk of an adverse outcome from participation in the trial.
* Likelihood of travel away from the study area.
* Positive malaria by blood smear at screening.
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Any other significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Ages: 5 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2023-08-27 (Actual); Study Completion 2023-08-27 (Actual)

PRIMARY OUTCOMES:
Safety of RH5.1-Matrix-M given in 3 doses in healthy Tanzanian adults and children naturally exposed to malaria as assessed by the occurrence of solicited symptoms. | Assessment of solicited symptoms in the first 7 days post vaccination
  Occurrence of solicited symptoms after each vaccination during a 7-day surveillance period.
Safety of RH5.1-Matrix-M given in 3 doses in healthy Tanzanian adults and children naturally exposed to malaria as assessed by the occurrence of unsolicited symptoms. | Assessment of unsolicited symptoms in the first 30 days post vaccination
  Occurrence of unsolicited symptoms after each vaccination during a 28-day surveillance period (day of vaccination and 28 subsequent days).
Safety of RH5.1-Matrix-M given in 3 doses in healthy Tanzanian adults and children naturally exposed to malaria as assessed by the occurrence of serious adverse events. | Assessment of SAEs until the end of the study (approx 2 years)
  Occurrence of serious adverse events throughout the study period.

SECONDARY OUTCOMES:
Anti-RH5 antibody concentration by ELISA | Through study completion (approx 2 years)
  Evaluation of the magnitude of antibody responses to RH5 in adults, children and infants residing in a malaria endemic country, as measured by ELISA
Growth inhibition activity of IgG from vaccinees on a panel of P. falciparum parasites | Through study completion (approx 2 years)
  Evaluation of the quality of antibody responses to RH5 in adults, children and infants residing in a malaria endemic country, as measured by an assay of growth inhibition activity on the vaccinees' sera
Avidity of anti-RH5 antibodies by ELISA and/or other assays (to be defined) | Through study completion (approx 2 years)
  Evaluation of the avidity of antibody responses to RH5 in adults, children and infants residing in a malaria endemic country, as measured by ELISA
Cellular immune responses to the RH5 by ELISpot assay and/or Flow cytommetry | Through study completion (approx 2 years)
  Evaluation of the magnitude and quality of cellular immune responses to PfRH5 in adults, children and infants residing in a malaria endemic country, by ELISpot assay and/or Flow cytommetry

CONTACTS AND LOCATIONS:
Overall Officials: Ally Olotu, Principal Investigator — Ifakara Health Institute
Locations (1):
- Ifakara Health Institute Clinical Trial Facility, Bagamoyo, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Study information will be made available through a repository. The information to be made available will be anonymized so that there is no link to participants and will include data on safety, immune responses and any other data generated from samples obtained in this study.
Supporting Information: Study Protocol
Time Frame: After publication of manuscripts related to the trial and for a minimum of 15 years from the end of the trial.
Access Criteria: Anonymized participant data will be made available when the trial is complete, upon requests directed to a corresponding author. Proposals will be reviewed and approved by the sponsor, investigators, and collaborators on the basis of scientific merit. After approval of a proposal, data can be shared through the secure online repository.

REFERENCES:
- [Derived] Silk SE, Kalinga WF, Salkeld J, Mtaka IM, Ahmed S, Milando F, Diouf A, Bundi CK, Balige N, Hassan O, Mkindi CG, Rwezaula S, Athumani T, Mswata S, Lilolime NS, Simon B, Msami H, Mohamed M, David DM, Mohammed L, Nyaulingo G, Mwalimu B, Juma O, Mwamlima TG, Sasamalo IA, Mkumbange RP, Kamage JJ, Barrett JR, King LDW, Hou MM, Pulido D, Carnrot C, Lawrie AM, Cowan RE, Nugent FL, Roberts R, Cho JS, Long CA, Nielsen CM, Miura K, Draper SJ, Olotu AI, Minassian AM. Blood-stage malaria vaccine candidate RH5.1/Matrix-M in healthy Tanzanian adults and children; an open-label, non-randomised, first-in-human, single-centre, phase 1b trial. Lancet Infect Dis. 2024 Oct;24(10):1105-1117. doi: 10.1016/S1473-3099(24)00312-8. Epub 2024 Jun 13. PMID 38880111
- [Derived] Mwamlima TG, Mwakasungula SM, Mkindi CG, Tambwe MM, Mswata SS, Mbwambo SG, Mboya MF, Draper SJ, Silk SE, Mpina MG, Vianney JM, Olotu AI. Understanding the role of serological and clinical data on assessing the dynamic of malaria transmission: a case study of Bagamoyo district, Tanzania. Pan Afr Med J. 2022 Oct 7;43:60. doi: 10.11604/pamj.2022.43.60.35779. eCollection 2022. PMID 36578806